CLINICAL TRIAL: NCT05278741
Title: Functional Evaluation After Breast Reconstruction With a Minimally Invasive Latissimus Dorsi Flap Following Radical Surgery for Breast Cancer.
Acronym: BREAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A03166-35
Record Dates: First submitted 2022-01-28; First posted 2022-03-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast; Latissimus dorsi flap
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, non-randomized interventional study in a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery for unilateral breast reconstruction (Experimental): Patients treated in oncological surgery at the Center Georges-François Leclerc (CGFL) in Dijon for unilateral breast reconstruction after therapeutic total mastectomy.
  Before the surgery, 2 questionnaires will be completed by patients : BREAST-Q and DASH. Also, the isokinetic test and EMG will be performed.
  After the surgery, 2 questionnaires will be completed at one month, 3 months, 6 months and 12 months. The Two tests will be performed at 3 months, 6 months and 12 months after the surgery.
  Interventions: Procedure: Surgery for unilateral breast reconstruction

INTERVENTIONS:
Procedure: Surgery for unilateral breast reconstruction — Before the surgery, patient will be completed two questionnaire DASH and BREAST-Q. Two tests will be performed (isokinetic test and EMG).
  After the surgery, at one month : 2 Questionnaires (DASH / BREAST-Q) will be performed At three months, six months and 12 months: 2 questionnaires + two tests will be perfomed

SUMMARY:
This study will quantify the muscle function after breast reconstruction using a minimally invasive latissimus dorsi flap.

The proposed measures (clinical, isokinetic, electrophysiology, function and quality of life questionnaires) allow a precise, multidisciplinary, objective evaluation of the capacity of the latissimus dorsi muscle before surgery, 3 months, 6 months and 12 months after surgery. A function deficit is expected (decreased moment of adduction and internal rotation) 3 months after surgery and a return to the preoperative state 6 months and 12 months after surgery.

ELIGIBILITY:
* Inclusion Criteria:

  1. Patient managed for unilateral MR (immediate or secondary) by MSLD after therapeutic mastectomy.
  2. Breast assessment (Mammography + ultrasound +/- breast MRI) normal dating less than 6 months
  3. Age between 18 and 80 years old
  4. Signature of free and informed consent
* Exclusion Criteria:

  1. Patient with metastasis or disease progression
  2. Patient whose general condition does not allow her to answer a questionnaire or perform physical and functional measurements (neurocognitive disorders and/or neuro-orthopedic disorders)
  3. Patient with a poor understanding of the French language
  4. Patient having presented a failure of a first breast reconstruction (failure of DIEP, prosthesis removal)
  5. Patient not eligible for MR secondary to cancer (prophylactic mastectomy) or for which the flap was intended to cover loss of substance and not reconstruction
  6. Patient with a history of contralateral MR (all techniques combined)
  7. Patient with a history of contralateral breast cancer
  8. Patient does not have internet access to be able to connect to the "Exolis" software

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Measurement of the muscular moment | During the 12 months post operation
  Measurement of the muscular moment of shoulder adduction preoperatively and at 3 months on an isokinetic dynamometer (Biodex®, New York, USA) at an adduction speed of 60 degrees per second during a maximal voluntary contraction

SECONDARY OUTCOMES:
Evaluation of muscle moments | During the 12 months post operation
  Evaluation of muscle moments, isokinetic measurements, performed on an isokinetic dynamometer (Biodex®, New York, USA) at different speeds (isometric, 30, 60 and 120 degrees per second) of adduction and internal rotation after flap surgery minimally invasive latissimus dorsi (measurements before surgery, at 3, 6 and 12 months)
Comparison of muscular moments | During the 12 months post operation
  Comparison of muscular moments on the operated and "healthy" sides at 3 months, 6 months and 12 months. Perfomed on an isokinetic dynamometer (Biodex®, New York, USA) at different speeds (isometric, 30, 60 and 120 degrees per second) of adduction and internal rotation after flap surgery minimally invasive latissimus dorsi
Calculation of adduction deficit | During the 12 months post operation
  Calculation of adduction deficit is defined as a relative difference of more than 5% compared to the measurement taken preoperatively. Patients who completed at least one physiotherapy session post-surgery and before 3 months will be compared to the others.
Measurement of surface electromyographic activity | During the 12 months post operation
  Measurement of surface electromyographic activity (sEMG) of the latissimus dorsi, teres major and pectoralis major muscles is measured before surgery, 3 months, 6 months and 12 months post-surgery
Functional clinical impact and quality of life | During the 12 months post operation
  Functional clinical impact and quality of life is evaluated by DASH questionnaire. These questionnaire will be administrated before surgery, 1 month, 3 months, 6 months and 12 months post-surgery.
  The DASH self-questionnaire is an upper limb function assessment scale. It offers the ability to perform 23 activities, the severity of the symptoms and optional sports or instrumental and professional activity.
Functional clinical impact and quality of life | During the 12 months post operation
  Functional clinical impact and quality of life is evaluated by BREAST-Q questionnaire. These questionnaire will be administrated before surgery, 1 month, 3 months, 6 months and 12 months post-surgery.
  The BREAST-Q questionnaire is a self-administered quality of life questionnaire assessing satisfaction after breast reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Clémentine CJ JANKOWSI, Dr, Principal Investigator — Centre Georges François Leclerc
Locations (1):
- Centre Georges-François Leclerc, Dijon, Côte d'Or, France